CLINICAL TRIAL: NCT02052440
Title: Preventing Alcohol Withdrawal Syndrome With Oral Baclofen: A Randomized, Placebo Controlled Trial
Brief Title: Preventing Alcohol Withdrawal Syndrome With Oral Baclofen
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Insufficient funding to complete with low enrollment rate
Sponsor: Denver Health and Hospital Authority (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 13-2883
Record Dates: First submitted 2014-01-30; First posted 2014-02-03 (Estimated); Results first posted 2018-03-27 (Actual); Last update posted 2018-05-23 (Actual); Status verified 2018-04

CONDITIONS: Alcohol Withdrawal Syndrome
MeSH Terms: interventions — Baclofen; Sugars

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Baclofen 10mg three times daily (Experimental): Baclofen 10mg by mouth three times daily
  Interventions: Drug: Baclofen
- Sugar Pill given three times daily (Placebo Comparator): Placebo sugar bill
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Baclofen — Treatment arm: baclofen 10mg tid
  Other Names: Baclofen 10mg will be given three times daily
  Arms: Baclofen 10mg three times daily
Drug: Placebo — Sugar pill by mouth three times daily
  Other Names: Sugar pill
  Arms: Sugar Pill given three times daily

SUMMARY:
Adult medical/surgical inpatient hospital care is more difficult and more expensive when complicated by alcohol dependency (AD), especially for patients who develop alcohol withdrawal syndrome (AWS). AWS can be mild, moderate or severe. The Severity of Ethanol Withdrawal Scale (SEWS) is tool used to assess severity and is the current standard of care for both monitoring and treating AWS at Denver Health. Moderate/severe AWS (i.e., SEWS ≥ 7) has important clinical implications and requires pharmacological treatment. At present, there are no safe and effective options for preventing AWS in at-risk inpatients. Baclofen is a GABA-B receptor agonist that has been used in the alleviation of spasticity in patients with multiple sclerosis since the 1970s. Baclofen has shown promise in the management of alcohol dependency in preclinical and clinical studies. We propose to examine baclofen in the prevention/amelioration of AWS in adult medical inpatients. The investigators hypothesize that Baclofen, as compared to placebo, will significantly reduce the number of adult inpatients with AD who will develop moderate/severe AWS (SEWS ≥ 7) when assessed at 72 hours after enrollment. Further the investigators hypothesize that Baclofen, as compared to placebo, will significantly reduce the need for symptom-triggered benzodiazepine administration during the 72 hours of hospitalization. These hypotheses will be tested in adult inpatients who are determined to be at risk for alcohol withdrawal and are subsequently placed on the SEWS monitoring and treatment protocol. These patients will be randomized to baclofen 10mg three times daily vs placebo.

DETAILED DESCRIPTION:
See Brief Summary. Patients will recieve standard of Care treatment and monitoring for ETOH withdrawl per our insitution wide SEWS protocol. They will then be randomized to recieve baclofen 10mg tid vs placebo tid for the course of their hospital stay or 7 days, whichever comes first.

ELIGIBILITY:
Inclusion Criteria:

* Adults age 21-100 admitted to medical floors at Denver Health
* Patients placed on SEWS protocol by admitting physicians (at risk for AWS).

Exclusion Criteria:

* Unable to provide informed consent
* Unable to take oral medications
* admitted for AWS or with SEWS score >7 at baseline
* no alcohol intake for ≥ 48 hours
* baclofen use at baseline
* baclofen sensitivity
* hospital discharge anticipated in within 48 hours
* pregnant or breast feeding (urine pregnancy test required of women of child-bearing potential
* other active drug dependence (except tobacco)
* taking a medication known to interact with baclofen.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2014-03-15; Primary Completion 2017-01-01 (Actual); Study Completion 2017-01-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel B Heppe, MD, Principal Investigator — Denver Health
Locations (1):
- Denver Health Hospital, Denver, Colorado, United States

IPD SHARING:
Plan to Share IPD: No
No plan to share individual patient data

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment and enrollment began March 1 2014 and terminated Jan 1 2017. Patients were enrolled after admission to general medical services at Denver Health Hospital.
Pre-assignment Details: Patients could be excluded if found to be pregnant prior to being assigned to study arm.
Period: Overall Study
Arm/Group | Baclofen 10mg Three Times Daily | Sugar Pill Given Three Times Daily
Started | 50 | 52
Completed | 50 | 51
Not Completed | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Baclofen 10mg Three Times Daily | Sugar Pill Given Three Times Daily | Total
Number analyzed (Participants) | 50 | 51 | 101
Age, Continuous [Mean (Standard Deviation); unit: Years] | 50 (10) | 51 (11) | 50 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 13 | 22
  Male | 41 | 38 | 79
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 4 | 3 | 7
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 7 | 11
  White | 41 | 41 | 82
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Prevention of Progression to Severe Alcohol Withdrawal as Assessed by Severity of Ethanol Withdrawal Score (SEWS).
Description: Prevention of progression to Severe Alcohol withdrawal as assessed by Severity of Ethanol Withdrawal Score (SEWS). A score of > 7 represents moderate alcohol withdrawal and a score > 12 severe alcohol withdrawal. Reported below as number of patients in each group progressing to moderate or severe alcohol withdrawal as assessed by SEWS score.
Time Frame: Within 72 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Baclofen 10mg Three Times Daily | Sugar Pill Given Three Times Daily
Number analyzed (Participants) | 50 | 51
Participants | 13 | 16

2. Secondary Outcome: Reduced Severity of Alcohol Withdrawal as Measured by Severity of Ethanol Withdrawal Score. .
Description: Severity of alcholol withdrawal will be assessed by monitoring SEWS scores in both baclofen and placebo group. This score is reported as a cumulative unit on scale ranging from 0 to 23. A value of 1-6 represents mild alcohol withdrawal, 7-12 moderate and >12 severe. Values will be measured 24 hours, 48 hours and 72 hours. A mean of these values was calculated.
Time Frame: Over 72 hours
Measure: Mean (Standard Deviation); unit: Unit on Scale
Arm/Group | Baclofen 10mg Three Times Daily | Sugar Pill Given Three Times Daily
Number analyzed (Participants) | 50 | 51
Unit on Scale
  Highest SEWS score at 24 hours | 6 (4) | 6 (4)
  Highest SEWS score at 48 hours | 4 (3) | 4 (4)
  Highest SEWS score at 72 hours | 2 (3) | 3 (3)

3. Secondary Outcome: Difference in Maximal Dose of Ethanol Withdrawal Symptom Driven Benzodiazepine Administration, as Assessed by SEWS Score, in Treatment Group When Compared to Placebo Group
Description: The null hypotheses of no difference in the maximum dose of inpatient symptom-triggered benzodiazepine therapy during the 72 hours following enrollment between those who receive baclofen and those who receive placebo. All maximum doses for each treatment arm given anytime between 0 and 72 hours were recorded and a mean calculated for each treatment arm.
Time Frame: 72 hours
Population: Maximum dose of symptom driven benzodiazepine
Measure: Mean (Standard Deviation); unit: Milligram of Diazepam
Arm/Group | Baclofen 10mg Three Times Daily | Sugar Pill Given Three Times Daily
Number analyzed (Participants) | 50 | 51
Milligram of Diazepam | 11 (2) | 12 (7)

4. Secondary Outcome: Difference in Cumulative Dose of Ethanol Withdrawal Symptom Driven Benzodiazepine Administration, as Assessed by SEWS Score, in Treatment Group Compared With Placebo Group.
Description: The null hypotheses of no difference in the cumulative inpatient dosages of symptom-triggered benzodiazepine therapy during the 72 hours following enrollment between those who receive baclofen and those who receive placebo. Total benzodiazepine administration received from 0 to 72 hours was summed for each patient in each arm. A mean of this cumulative dose was then calculated for each arm and is reported below.
Time Frame: 72 hours
Population: Cumulative dose of symptom driven benzodiazepine
Measure: Mean (Standard Deviation); unit: Milligram of Diazepam
Arm/Group | Baclofen 10mg Three Times Daily | Sugar Pill Given Three Times Daily
Number analyzed (Participants) | 50 | 51
Milligram of Diazepam | 66 (51) | 85 (63)

ADVERSE EVENTS:
Time Frame: While subject inpatient and enrolled in study until time of discharge or maximum 96 hours, whichever came first.
Description: Study personnel checked with nursing and treatment teams daily to monitor for adverse events
Arm/Group | Baclofen 10mg Three Times Daily | Sugar Pill Given Three Times Daily
All-Cause Mortality (participants affected / at risk) | 0/50 | 0/51
Serious Adverse Events (participants affected / at risk) | 0/50 | 0/51
Other Adverse Events (participants affected / at risk) | 1/50 | 0/51
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Baclofen 10mg Three Times Daily (N=50) | Sugar Pill Given Three Times Daily (N=51)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — Patient developed rash 36 hours following initiation of study medication. Study medication was discontinued and rash improved and patient discharged

LIMITATIONS AND CAVEATS:
The number of patients enrolled was less than was needed based on our sample size estimation due to termination of study secondary to funding limitations. This study was performed at a single, university-affiliated public safety net hospital.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No